CLINICAL TRIAL: NCT03787498
Title: A Phase 1b Dose-escalation Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of PLX2853 in Subjects With Relapsed or Refractory Acute Myeloid Leukemia or High-risk Myelodysplastic Syndrome
Brief Title: A Study of PLX2853 in Relapsed or Refractory Acute Myeloid Leukemia or High Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Opna Bio LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLX124-02
Record Dates: First submitted 2018-12-23; First posted 2018-12-26 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Relapsed Acute Myeloid Leukemia (AML); Refractory Acute Myeloid Leukemia (AML); High-risk Myelodysplastic Syndrome (MDS)
Keywords: PLX2853; Acute Myeloid Leukemia; AML; Myelodysplastic Syndrome; MDS; Hematologic Malignancy; Blood Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PLX2853 (Experimental): Approximately 30 subjects will be enrolled as part of dose escalation to identify the MTD/RP2D of PLX2853. Up to 6 additional subjects may be enrolled at the MTD/RP2D to further characterize the PK and PDy of PLX2853.
  Interventions: Drug: PLX2853

INTERVENTIONS:
Drug: PLX2853 — Tablets

SUMMARY:
The purpose of this research study is to evaluate safety, pharmacokinetics, pharmacodynamics and preliminary efficacy of the investigational drug PLX2853 in subjects with Relapsed or Refractory Acute Myeloid Leukemia or High-risk Myelodysplastic Syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of one of the following myeloid malignancies, based on the 2016 revision of the World Health Organization classification:

   A. Relapsed or refractory AML.

   I. Subjects must have received no more than 3 prior induction therapies and have no standard therapeutic option that is expected to result in a clinical benefit.

   B. Relapsed or refractory MDS.

   I. Subjects must have high-risk disease (intermediate or greater disease according to the revised International Prognostic Scoring System [IPSS-R]).

   II. Subjects must have received no more than 3 prior therapies, 1 of which must have included a hypomethylating agent such as azacytidine or decitabine.

   III. Subjects must have no standard therapeutic option that is expected to result in a clinical benefit.
2. Age ≥18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
4. Life expectancy of ≥3 months in the judgment of the investigator.
5. Adequate renal, hepatic, and coagulation parameters:

   A. Measured or calculated (Cockcroft-Gault formula) creatinine clearance (CrCl) ≥60 mL/min.

   B. Total bilirubin ≤1.5 × ULN unless due to Gilbert's syndrome.

   C. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN.

   D. Prothrombin time or international normalized ratio ≤1.5 × ULN.

   E. Activated partial thromboplastin time ≤1.5 × ULN.
6. Women of child-bearing potential must have a negative pregnancy test at Screening and must agree to use an effective form of contraception from the time of the negative pregnancy test to 90 days after the last dose of study drug. Effective forms of contraception include abstinence, hormonal contraception in conjunction with a barrier method, or a double barrier method. Women of non-child-bearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year.
7. Fertile men must agree to use an effective method of birth control during the study and for 90 days after the last dose of study drug.
8. Resolution (to ≤Grade 1 or baseline) of all significant toxicity associated with prior cancer therapy prior to study drug initiation. (Grade 2 alopecia or residual Grade 2 peripheral neuropathy is allowed.)
9. Willingness and ability to provide written informed consent prior to any study-related procedures and to comply with all study requirements.

Exclusion Criteria:

1. Prior treatment with a bromodomain inhibitor.
2. Any one of the following therapies:

   A. Stem cell transplantation within 90 days of study drug initiation;

   B. Active immunosuppressive therapy for graft-versus-host disease (GVHD);

   C. GVHD prophylaxis within 2 weeks of study drug initiation.
3. Known uncontrolled fungal, bacterial, and/or viral infection ≥Grade 2.
4. Uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia.
5. Active symptomatic central nervous system involvement of AML. (Individuals who have had leptomeningeal disease that was effectively treated are eligible.)
6. A diagnosis of acute promyelocytic leukemia or chronic myeloid leukemia in blast crisis.
7. Known or suspected allergy to the study drug or any agent given in association with this trial.
8. Women who are either pregnant or breast feeding.
9. Clinically significant cardiac disease.
10. Inability to take oral medication or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the Investigator, would preclude adequate absorption.
11. Individuals who are known to be infected with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV) or are known carriers of HBV or HCV. Individuals who are positive for HCV antibody must be negative for HCV RNA by polymerase chain reaction (PCR) to be eligible. Individuals with occult or prior HBV infection (defined as being seropositive for total hepatitis B core antibody and seronegative for hepatitis B surface antigen) may be included if HBV DNA is undetectable. These individuals must be willing to undergo additional testing per local standard of care.
12. Active second malignancy with the exception of any of the following:

    * Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer;
    * Adequately treated Stage I cancer from which the subject is currently in remission and has been in remission for ≥2 years;
    * Low-risk prostate cancer with Gleason score <7 and prostate-specific antigen <10 ng/mL;
    * Any other cancer from which the patient has been disease-free for ≥3 years.
13. Major surgery or significant injury within the 14-day period prior to study drug initiation.
14. Anti-cancer therapy in the period immediately preceding study drug initiation.
15. Any other medical, psychological, familial, sociologic, or geographic condition that, in the judgement of the investigator, would potentially hamper compliance with the study protocol or interfere with the study endpoints or the subject's ability to participate in the study.
16. Participation in any other therapeutic clinical study. (Participation in observational or registry trials is allowed.)
17. Individuals who are on active anticoagulation therapy (e.g., warfarin, factor Xa inhibitors, thrombin inhibitors, heparin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | First dose of study drug through at least 30 days after end of treatment
Area under the concentration-time curve (AUC) of PLX2853 | From first dose of PLX2853 up to 30 days after end of treatment
Maximum observed concentration (Cmax) of PLX2853 | From first dose of PLX2853 up to 30 days after end of treatment
Time to peak concentration (Tmax) of PLX2853 | From first dose of PLX2853 up to 30 days after end of treatment
Half life (t1/2) of PLX2853 | From first dose of PLX2853 up to 30 days after end of treatment
Terminal elimination rate constant (Kel) | From first dose of PLX2853 up to 30 days after end of treatment
Number of participants who experience dose limiting toxicity as defined in the protocol | up to 18 months
  Dose escalation will be guided by a modified continuous reassessment method (mCRM) using a Bayesian logistic regression model that follows the escalation with overdose control (EWOC) principle. In this method, a decision to escalate to the next dose level is based on a review of all subjects who have completed the DLT observation period.

SECONDARY OUTCOMES:
Overall complete remission (OCR) rate | From the first dose of study drug until the date of documented best response to treatment, assessed up to 18 months
  AML - Complete Remission (CR) + CR with incomplete hematological recovery (CRi); MDS - CR
Overall response rate (ORR) | From the first dose of study drug until the date of documented response to treatment, assessed up to 18 months
  AML - Complete Remission (CR) + CR with incomplete hematologic recovery (CRi) + Partial Remission (PR); MDS - CR + PR
Duration of response (DOR) | DOR defined as the time from the initial objective response to disease progression or death, whichever occurs first, assessed up to 18 months
Event-free survival (EFS) | EFS time is defined as the time from the first dose of PLX2853 to treatment failure, relapse after initial response or death from any cause, assessed up to 18 months.
Progression-free survival (PFS) | PFS time is defined as the time from the first dose of PLX2853 to disease progression or death, whichever occurs first, assessed up to 18 months.
Overall survival (OS) | From the first dose of study drug until the date of death from any cause, assessed up to 18 months.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Northside Hospital, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer At Johns Hopkins, Baltimore, Maryland
  - NewYork-Presbyterian / Weill Cornell Medical Center, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Texas MD Anderson Cancer Center, Houston, Texas